CLINICAL TRIAL: NCT00962806
Title: Intensive Exercise to Improve Mitochondrial Dysfunction in Pediatric Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amy Fleischman, MD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK084118; Partners IRB: 2009P-000173
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Pediatric Obesity; Insulin Resistance; Mitochondrial Dysfunction
Keywords: Pediatric obesity; Insulin resistance; Diabetes; Mitochondria
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Mitochondrial Diseases; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Active Comparator): 8 week intensive exercise group
  Interventions: Behavioral: Exercise
- Control Lifestyle counseling (Other): Lifestyle counseling without intensive exercise
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Exercise — 8 weeks of intensive exercise, 60-90 minutes 3 days each week
  Arms: Exercise
Behavioral: Lifestyle counseling — Baseline and final visit dietary and activity advice and weekly healthy lifestyle messages
  Arms: Control Lifestyle counseling

SUMMARY:
Obesity and type 2 diabetes are occurring at epidemic rates in the United States and worldwide. The global burden of diabetes is estimated to double over the next 25 years. Obese children are at risk for the development of insulin resistance, relative insulin deficiency and type 2 diabetes mellitus (DM). The prevention of type 2 DM is hindered by the lack of a non-invasive predictive test, knowledge as to individual risk and effective preventative measures. There is increasing evidence that alterations in mitochondria contribute to the development of diabetes in humans. Therefore, it is important to explore mitochondrial dysfunction as a potential predictor of diabetes in children and a potential target for prevention. The aims of the proposed protocol are to determine whether an intensive exercise intervention can improve mitochondrial function in children identified as having mitochondrial dysfunction and insulin resistance. The use of a non-invasive imaging technique will allow for a functional in vivo assessment of mitochondrial activity. The investigators propose the investigation of an intensive exercise protocol designed to improve mitochondrial function in children who are insulin resistant and have documented mitochondrial dysfunction by magnetic resonance spectroscopy. The study is designed to investigate the plasticity of abnormal mitochondrial function in high risk children. In summary, the proposed projects will investigate mitochondrial function as a non-invasive predictive marker for the development of insulin resistance and type 2 diabetes mellitus in children and attempt to modify mitochondrial function with an intensive exercise intervention. The study of mitochondrial dysfunction in children may both identify those at risk for disease and provide a molecular therapeutic target for prevention and treatment.

The investigators hypothesize that children with insulin resistance and mitochondrial dysfunction who are randomized to intensive exercise versus standard lifestyle advice will show improvement in mitochondrial function and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys ages 10 to 18 years old
* Body mass index more than 95th percentile for age and gender
* Insulin resistance based on:

  * Fasting parameters: Fasting insulin level, HOMA IR
  * Oral glucose tolerance testing
* Mitochondrial function > 1 median for normal based on control cohort

Exclusion Criteria:

* Underlying medical problem with potential to affect growth, pubertal development or glucose homeostasis
* Chronic medical therapy with glucocorticoids, growth hormone, estrogen, progesterone, testosterone, or other medications with the potential to alter growth, pubertal development or glucose homeostasis within the proceeding 6 months
* Personal history of DM
* Inability to have MRI scan performed due to metal prosthesis or implant

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determine whether intensive exercise improves mitochondrial function by P31 MRS and mitochondrial number by peripheral blood analyses. | 2 year

SECONDARY OUTCOMES:
Determine whether intensive exercise improves metabolic parameters and glucose metabolism. | 2 years
Determine whether intensive exercise improves body composition, by DXA, and intramyocellular fat content, by 1H MRS. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States